CLINICAL TRIAL: NCT04826835
Title: A Prehabilitation Program to Boost Postoperative Functional Capacity in Surgical Lung Cancer Patients: a Randomized Controlled Trial
Brief Title: A Prehabilitation Program to Boost Postoperative Functional Capacity in Surgical Lung Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Chia-Chin Lin, Professor and Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW 19-214
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer
Keywords: Prehabilitation; Physical activity; Lung resection; Functional capacity
MeSH Terms: conditions — Lung Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation intervention (Experimental): Participants in the intervention group will follow a 2-week prehabilitation program before lung resection.
  Interventions: Behavioral: Prehabilitation intervention
- Health education control (Active Comparator): Participants in the control group will receive health education classes during 2 weeks before lung resection.
  Interventions: Behavioral: Health education control

INTERVENTIONS:
Behavioral: Prehabilitation intervention — Participants will:
  * Receive four supervised exercise classes (twice per week for two weeks) one-to-one by an exercise specialist;
  * Practice six sessions of home-based exercise (three times per week for two weeks);
  * Practice unsupervised respiratory muscle training at home (twice daily for two weeks);
  * Receive usual care.
  Arms: Prehabilitation intervention
Behavioral: Health education control — Participants will:
  * Receive four recorded health education talks (twice per week for two weeks)
  * Receive a brief health education booklet on dietary education for chronic lung conditions, preoperative preparation, and postoperative recovery
  * Receive usual care.
  Arms: Health education control

SUMMARY:
This research study is evaluating a prehabiliation intervention designed to improve postoperative functional capacity (measured by 6-minure walking distance) in individuals undergoing lung resection for cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed of stage I, II, or IIIA Non-small-cell lung carcinoma (NSCLC) diagnosis, with or without pre-operative histologic confirmation
2. Patients scheduled to undergo lung resection surgery at least two weeks from recruitment
3. Patients with a Eastern Cooperative Oncology Group (ECOG) score of 0 or 1 at recruitment
4. Patients with no evidence of recurrent or progressive disease
5. Patients aged 45-80 years
6. Patients able to communicate in Cantonese, Mandarin, or English
7. Patients is absence of any cognitive impairment
8. Patients with a score of 6 minutes walking test (6MWT) ≤ 500 meters at baseline. [rationale: a threshold value of 500 meters preoperative 6MWT predicts a higher risk of postoperative complications and prolonged LOS after lung resection]
9. Engagement in less than 150 minutes of moderate aerobic activity per week in the past 3 months

Exclusion Criteria:

1. Patients who had engaged in at least 150 minutes of moderate aerobic activity or 75 minutes of vigorous aerobic activity per week in the past three months
2. Presence of another concurrent, actively treated malignancy
3. Presence of chronic obstructive pulmonary disease
4. Presence of significant comorbidities that impede ability to engage in exercise, such as congestive heart failure, orthopedic disorders of the lower limbs, respiratory failure, or the need for portable oxygen therapy for activities of daily living
5. Not having a smart device to receive WhatsApp messages

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline 6-minute walking distance from baseline to 3-month post-surgery | Baseline; 3-month post-surgery

SECONDARY OUTCOMES:
Change from baseline 6-minute walking distance at post-intervention | Baseline; 2 weeks (post-intervention)
Change from baseline 6-minute walking distance at 1-month post-surgery | Baseline; 1-months post-surgery
Length of postoperative hospital stay | 1-month post-surgery
Postoperative complication | 1-month post-surgery
Change from baseline functional assessment of cancer treatment - Lung (FACT-L) at post-intervention | Baseline; 2 weeks (post-intervention)
Change from baseline functional assessment of cancer treatment - Lung (FACT-L) at 1-month post-surgery | Baseline; 2 weeks (post-intervention); 1-month post-surgery
Change from baseline functional assessment of cancer treatment - Lung (FACT-L) at 3-months post-surgery | Baseline; 3-month post-surgery
Change from baseline international physical activity questionnaire (IPAQ) at post-intervention | Baseline; 2 weeks (post-intervention)
Change from baseline international physical activity questionnaire (IPAQ) at 1-month post-surgery | Baseline; 1-month post-surgery
Change from baseline international physical activity questionnaire (IPAQ) at 3-month post-surgery | Baseline; 3-month post-surgery
Change from baseline daily step count measured by pedometer at post-intervention | Baseline; 2 weeks (post-intervention)
Change from baseline daily step count measured by pedometer at 1-month post-surgery | Baseline; 1-month post-surgery
Change from baseline daily step count measured by pedometer at 3-month post-surgery | Baseline; 3-month post-surgery
Health-related quality of life for the cost-effectiveness analysis (EuroQol- 5 Dimension, EQ-5D-5L) | Baseline; 2 weeks (post-intervention); 1-month post-surgery; 3-month post-surgery
Health-related quality of life for the cost-effectiveness analysis (EuroQol-Visual Analog Score, EQ-VAS) | Baseline; 2 weeks (post-intervention); 1-month post-surgery; 3-month post-surgery
Physical activity self-efficacy (9-item Self-Efficacy for Exercise, SEE) | Baseline; 2 weeks (post-intervention); 1-month post-surgery; 3-month post-surgery
Financial toxicity (COmprehensive Score for financial Toxicity, COST questionnaire) | Baseline; 3-month post-surgery
Return to work (investigator-designed questionnaire) | 3-month post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No